CLINICAL TRIAL: NCT01478113
Title: Stimulant Enhancement of Well-Being Therapy for Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution and was no funding to continue study.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Maren Nyer, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011P002148; 2011D002171 (Other Grant/Funding Number: InfoED ID: Kaplen Fellowship and Livingston Award)
Record Dates: First submitted 2011-09-26; First posted 2011-11-23 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Therapy; Medication study; Depression; Therapy study
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — SLI381; Adderall

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- WBT + amphetamine/dextroamphetamine (Active Comparator): In the active group, participants will receive treatment with Well-being therapy and amphetamine-dextroamphetamine.
  Interventions: Drug: Amphetamine/dextroamphetamine; Behavioral: Well-being therapy
- WBT + placebo (Placebo Comparator): In the placebo group, participants will receive treatment with Well-being therapy and pill placebo.
  Interventions: Drug: Placebo; Behavioral: Well-being therapy

INTERVENTIONS:
Drug: Amphetamine/dextroamphetamine — The amphetamine/dextroamphetamine will be in a pill formulation. The dosage of the amphetamine/dextroamphetamine will be flexibly adjusted up or down by a study clinician based on the participant's response. Dose ranges will be 1-3 pills (placebo or 5 mg amphetamine) in the morning and 1-3 pills (placebo or 5 mg amphetamine) at noon.
  Other Names: Adderall; Adderall XR
  Arms: WBT + amphetamine/dextroamphetamine
Drug: Placebo — The placebo will match the dextroamphetamine in form, dosage, frequency, and duration.
  Other Names: Sugar-pill
  Arms: WBT + placebo
Behavioral: Well-being therapy — Therapy sessions will last between 30-50 minutes. The sessions will take place at every visit after the screening visit.
  Other Names: WBT

SUMMARY:
This study aims to identify a novel enhancement strategy for residual symptoms of major depressive disorder (MDD) Dopamine (DA) has been viewed as a "pleasure neurotransmitter" for over 30 years. Yet recent data from animal and human studies suggest that dopamine has greater effects on "wanting" than on "liking." Therefore, the investigators of this study have hypothesized that amphetamine/d-amphetamine (AMPH), a medication which increases dopamine transmission in the reward centers of the brain, may have a more powerful antidepressant effect in combination with well-being therapy (WBT), a specific type of cognitive-behavioral therapy, which helps individuals with depression to increase their contact with natural rewards and decrease reward-interfering thoughts.

The investigators will test their hypothesis by randomizing 40 individuals with residual symptoms of depression, already taking an antidepressant that affects serotonin (e.g. Prozac, Paxil), to 8 weeks of treatment with either WBT in combination with AMPH, or WBT with pill placebo. The effectiveness of each treatment will be measured using a reliable scale, called the Hamilton Depression Rating Scale.

The investigators have also hypothesized that people assigned to the stimulant/WBT group will have greater improvements in functioning, well-being, and positive affectivity than those the people assigned to the WBT/placebo group.

DETAILED DESCRIPTION:
The study will have 11 visits occur over 8 weeks with study visits scheduled weekly or biweekly.

Detailed Description:

The study visit occurrences are as follows:

1. Week 0- Screening Visit
2. Week 1- Baseline Visit
3. Week 2- one phone visit and one clinic visit in one week
4. Week 3- one phone visit and one clinic visit in one week
5. Week 4- one visit in one week
6. Week 5- one visit in one week
7. Week 6- one visit in one week
8. Week 7- one visit in one week
9. Week 8- one visit in one week

WBT description Four licensed therapists, who have been trained and certified in WBT, will provide weekly sessions of 30 to 50 minutes in duration. Therapists will follow the procedures outlined in the WBT manual. The initial sessions (weeks 0-2) will be focused on identifying and contextualizing episodes of well-being. The intermediate sessions (weeks 3-5) will be focused on modifying cognitions and behaviors, which lead to premature interruption of well-being, and optimizing cognitions and behaviors, which have been idiographically linked to enhanced well-being. Final sessions (weeks 6-8) will apply the Psychological Well-Being scales (PWB) to refine treatment according to Ryff's dimensions of well-being. Additional principles and techniques of WBT include reappraisal, mood-charting, scheduling of activities, shaping, problem-solving, and assertiveness training.

Medication Schedule Participants will receive treatment with the stimulant, amphetamine/d-amphetamine, or matched placebo.

Participants will start at 1 pill (placebo or 5 mg amphetamine/d-amphetamine) in the morning and 1 pill (placebo or 5 mg amphetamine/d-amphetamine) at noon. The treatment will then be flexibly adjusted up or down by a study clinician based on participant's response. Dose ranges will be 1-3 pills (placebo or 5 mg amphetamine) in the morning and 1-3 pills (placebo or 5 mg amphetamine) at noon.

ELIGIBILITY:
Inclusion Criteria

1. Outpatients between 18 and 60 years of age.
2. Experiencing residual symptoms after 8 weeks of SSRI therapy, with at least 4 weeks at a stable dose of the current agent prior to randomization.
3. Fulfillment of DSM-IV diagnostic criteria for MDD during the present episode of illness with continuing residual symptoms.
4. A score of 14 to 26 on the 31-item Hamilton Depression Rating Scale (HAM-D-31) at screening and randomization.
5. A Clinical Global Impression of Severity (CGI-S) score of 3 or 4 at screening and randomization.

Exclusion Criteria

1. Treatment within 4 weeks of randomization with any non-SSRI antidepressant, antipsychotic, mood stabilizer, standing benzodiazepine, stimulant, or stimulant-like agent.

   1. Allowed exception 1: Concomitant benzodiazepines, at a stable dose, that have been taken for at least one year with no history of abuse.
   2. Allowed exception 2: Effexor, duloxetine (Cymbalta) or milnacipran (Savella) can serve as main SSRI treatment.
   3. Allowed exception 3: Combinations of SSRIs (ex. Zoloft & Lexapro concomitantly) are acceptable as main SSRI treatment.
2. If a subject endorses "yes" or "agree" of any item from 12 to 23 on the CHRT, it would indicate active suicidality and would be exclusionary.
3. Significant suicide risk.
4. Current treatment-resistant episode of MDD.
5. A primary diagnosis of an Axis I disorder other than MDD.
6. History of a psychotic disorder, dysthymia, antisocial personality disorder, BPD, or mental retardation.
7. History of a substance use disorder, with the exception of nicotine dependence, within 12 months prior to screening.
8. History of stimulant abuse, prescription drug abuse, and eating disorders.
9. Initial insomnia at screening that is not adequately controlled by medications. Subjects with recent history of unstable insomnia as defined by active or poorly controlled symptoms of insomnia within the past 1 month will be excluded.
10. Co-morbid medical conditions including a structural heart defect or rhythm abnormality that might be exacerbated by stimulant therapy; hypertension as measured by a resting sitting systolic blood pressure of > 149mmHg or diastolic blood pressure > 95mmHg; tachycardia as measured by a sitting pulse rate of >100 bpm or <50 bpm after resting for 5 minutes.
11. Allergy, hypersensitivity, intolerance, or history of non-responsivity to stimulant medications.
12. History of non-responsivity to CBT or well-being therapy.
13. Women who are pregnant or breastfeeding.
14. Glaucoma or hyperthyroidism
15. Current concomitant therapy is only permitted if it is supportive therapy (not specifically CBT) and has been ongoing for at least one year. However, if a subject has been in therapy for less than one year and wishes to discontinue or take a hiatus from their current therapy before coming in for a screening visit, this will be allowed. Additionally, subjects may not enter into other talk therapies for the duration of this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital and Harvard Medical School
Locations (1):
- Depression Clinical and Research Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available.

RESULTS

PARTICIPANT FLOW:
Groups:
- Well-being Therapy With Amphetamine/Dextroamphetamine: In the active group, participants will receive treatment with Well-being therapy and amphetamine-dextroamphetamine.
  Amphetamine-dextroamphetamine (AMPH): The amphetamine-dextroamphetamine will be in a pill formulation. The dosage of the amphetamine-dextroamphetamine will be flexibly adjusted up or down by a study clinician based on the participant's response. Dose ranges will be 1-3 pills (placebo or 5 mg amphetamine) in the morning and 1-3 pills (placebo or 5 mg amphetamine) at noon.
  Well-being therapy: Therapy sessions will last between 30-50 minutes. The sessions will take place at every visit after the screening visit.
- Well-being Therapy With Placebo: In the placebo group, participants will receive treatment with Well-being therapy and pill placebo.
  Placebo: The placebo will match the dextroamphetamine in form, dosage, frequency, and duration.
  Well-being therapy: Therapy sessions will last between 30-50 minutes. The sessions will take place at every visit after the screening visit.
Period: Overall Study
Arm/Group | Well-being Therapy With Amphetamine/Dextroamphetamine | Well-being Therapy With Placebo
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Well-being Therapy With Amphetamine/Dextroamphetamine | Well-being Therapy With Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 50 [45 to 55] | 54 [53 to 55] | 52 [45 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton-Depression Rating Scale(SIGH-D)-17 Items
Description: Comparison between the 2 groups of the percentage of subjects in remission, as defined by a HAM-D-17 score of < 8 at endpoint visit 11/week 8 of treatment, or early termination visit.
Time Frame: Baseline and visit 11/week 8 of treatment, or between baseline and early termination visit.
Population: not able to analyze due to small sample size
Arm/Group | Well-being Therapy With Amphetamine/Dextroamphetamine | Well-being Therapy With Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Hamilton-Depression Rating Scale(SIGH-D)-31 Item
Description: Comparison between the 2 groups of the percentage of participants who have responded to the treatment (response is defined here as a 50% or greater improvement on the HAM-D-31 score) between Baseline and Visit 11 or Early Termination Visit.
Time Frame: Baseline to Visit 11 (which is week 8 of treatment) or Early Termination Visit.
Population: not able to analyze due to small sample size
Arm/Group | WBT + Amphetamine/Dextroamphetamine | WBT + Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Psychological Well-being Scale (PWB)
Description: Well-being improvement: Comparison between the 2 groups of changes on the PWB at Baseline and Visit 11/Early Termination.
Time Frame: Baseline to Visit 11 (which is 8 weeks of treatment) or Early Termination Visit.
Population: not able to analyze due to small sample size
Arm/Group | Well-being Therapy With Amphetamine/Dextroamphetamine | Well-being Therapy With Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in the Snaith-Hamilton Pleasure Scale (SHAPS)
Description: Improvement of anhedonia: Comparison between the 2 groups of changes on the SHAPS at Baseline and Visit 11/Early Termination.
Time Frame: Baseline to Visit 11 (which is 8 weeks of treatment) or Early Termination Visit.
Population: not able to analyze due to small sample size
Arm/Group | WBT + Amphetamine/Dextroamphetamine | WBT + Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Behavioral Inhibition/Activation Scale (BIS/BAS)
Description: Improvement of deficits in behavioral activation: Comparison between the 2 groups of changes on the BIS/BAS at Baseline and Visit 11/Early Termination.
Time Frame: Baseline to Visit 11 (which is 8 weeks of treatment) or Early Termination Visit.
Population: not able to analyze due to small sample size
Arm/Group | Well-being Therapy With Amphetamine/Dextroamphetamine | Well-being Therapy With Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Positive and Negative Affective Scale (PANAS)
Description: Improvement of deficits in positive affectivity: Comparison between the 2 groups of changes on the PANAS at Baseline and Visit 11/Early Termination.
Time Frame: Baseline to Visit 11 (which is 8 weeks of treatment) or Early Termination Visit.
Population: not able to analyze due to small sample size
Arm/Group | Well-being Therapy With Amphetamine/Dextroamphetamine | Well-being Therapy With Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Functioning on Short Form-12(SF-12)
Description: Functional improvement: Comparison between the 2 groups of changes on the SF-12 scale at Baseline and Visit 11/Early termination visit.
Time Frame: Baseline to Visit 11 (which is 8 weeks of treatment) or Early Termination Visit.
Population: not able to analyze due to small sample size
Arm/Group | Well-being Therapy With Amphetamine/Dextroamphetamine | Well-being Therapy With Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Over the course of participant enrollment in the study (at each visit between Baseline and Visit 11), the total duration of which was 8 weeks.
Arm/Group | Well-being Therapy With Amphetamine/Dextroamphetamine | Well-being Therapy With Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Well-being Therapy With Amphetamine/Dextroamphetamine (N=2) | Well-being Therapy With Placebo (N=2)
Insomnia and Headache (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was shut down due to original PI leaving the institution and due to lack of continued funding. As such, we were not able to enroll a sufficient number of patients to analyze data/answer study hypothesis/achieve study aims.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes